CLINICAL TRIAL: NCT07039825
Title: Abdominal Aortic Aneurysm CTA Cohort Study (AAA-CTA Registry)
Brief Title: AAA-CTA Cohort Registry
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AAA-CTA cohort
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm; Image
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Computed tomography angiography — The results of computed tomography angiography on abdominal aortic aneurysm are collected.

SUMMARY:
The aim of this study is to investigate the measurement of abdominal aortic aneurysm by computed tomography angiography. The research will collected the results of computed tomography angiography from inpatient, emergency, and outpatient populations with abdominal aortic aneurysm.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is a life-threatening vascular disorder characterized by irreversible dilation of the abdominal aorta, posing a significant risk of rupture and catastrophic hemorrhage, with mortality rates reaching 65-85% upon rupture. Given the often asymptomatic nature of AAA until rupture, early detection and precise monitoring are critical to prevent fatal outcomes, underscoring the urgent need for reliable diagnostic tools.

Computed tomography angiography (CTA) has emerged as a gold-standard non-invasive imaging technique, offering high-resolution visualization of AAA morphology, including aneurysm diameter, wall thickness, thrombus formation, and spatial relationship to adjacent structures, which are essential for accurate diagnosis, rupture risk stratification, and surgical planning.

This study aims to investigate the precision and clinical utility of CTA in AAA measurement, with the potential to optimize screening protocols, improve intervention timing, and ultimately reduce AAA-related mortality.

By establishing standardized CTA-based assessment criteria, this research may contribute to enhanced diagnostic workflows, better patient risk stratification, and more personalized treatment strategies, thereby addressing a critical gap in vascular disease management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with abdominal aortic aneurysm who visited the study hospital.
2. Patients included should have computed tomography angiography data.

Exclusion Criteria:

1. Patients who declined participation, cases with incomplete or missing clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysm undergoing computed tomography angiography
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximal abdominal aortic diameter | 1 month
  The images of computed tomography angiography on abdominal aortic aneurysm are collected and the maximal diameter of abdominal artery is measured by medical specialists.

SECONDARY OUTCOMES:
Rupture | 1 month
  The images of computed tomography angiography on abdominal aortic aneurysm are collected and the rupture of AAA is judged by medical specialists.
Mortality | 1 month
  The death of AAA patients is recorded and mortality is calculated.
Other characteristics of AAA morphology | 1 month
  Through CTA images, the existence of ulcer, mural thrombus is judged, and the length of AAA is measured by medical specialists.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided